CLINICAL TRIAL: NCT06981052
Title: Prospective Evaluation of an Endoscopic Ultrasound (EUS)-Based Artificial Intelligence to Assist in the Deployment of Lumen Apposing Metal Stents for Gallbladder Drainage
Acronym: EUS-AI GBD
Status: Recruiting | Type: Observational
Sponsor: University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, Neil Marya, Assistant Clinical Professor of Medicine, University of Massachusetts, Worcester
Other Study IDs: H00020934
Record Dates: First submitted 2025-04-24; First posted 2025-05-20 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-05

CONDITIONS: Cholecystitis
MeSH Terms: conditions — Cholecystitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with gallbladders undergoing AI evaluation for stent deployment

SUMMARY:
Lumen apposing metal stents are now being used to help patients who suffer from cholecystitis (infection of the gallbladder), especially in cases where patients are not candidates for surgery. Lumen apposing metal stents are effective for draining the gallbladder, however, placement is technically challenging. Scientists have developed an artificial intelligence to aid doctors in the deployment of these stents into the gallbladder. The aim of this study is test the performance of an artificial intelligence in providing physicians accurate information for gallbladder drainage.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Anticipation that patient may undergo endoscopic ultrasound
* Gallbladder present

Exclusion Criteria:

* Cholecystectomy
* No indication for endoscopic ultrasound

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing endoscopic ultrasound who have a gallbladder present
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2025-05-12 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Accuracy of the EUS AI system in providing a recommendation (i.e. whether it is safe or not to drain the gallbladder) | Day 1
  An expert endoscopist will perform the endoscopic ultrasound procedure. When the gallbladder comes into view the expert will comment as to whether they believe that the gallbladder is safe to drain. The expert will be blinded to the AI computers interpretation of the view of the gallbladder. A second observer will record what the AI recommended at the time of the blinded expert. The expert will be considered the "gold standard" and the outcome will be accuracy of the AI in mimicking the experts recommendations.

CONTACTS AND LOCATIONS:
Locations (1):
- UMass Chan Medical School/Umass Memorial Health Care, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Other researchers can reach out to UMass Chan to obtain deidentified data on a case-by-case basis.
Supporting Information: Study Protocol, SAP